CLINICAL TRIAL: NCT03090945
Title: Pediatric Acute Bleeding Registry: Identification of Clinical, Laboratory and Endoscopic Risk Factors Associated With Pediatric Upper Gastrointestinal Bleeding
Brief Title: Pediatric Acute Gastrointestinal Bleeding Registry
Acronym: TRIAGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: Baylor College of Medicine (Other); Children's Medical Center Dallas (Other); University of Massachusetts, Worcester (Other); Children's Hospital of Philadelphia (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Michael A. Manfredi, MD, Assistant Professor of Pediatrics, Harvard Medical School, Boston Children's Hospital
Other Study IDs: P00021336
Record Dates: First submitted 2017-03-20; First posted 2017-03-27 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Upper Gastrointestinal Bleeding; Gastro Intestinal Bleeding
Keywords: Endoscopy; GI Bleeding; Pediatrics; Upper Gastrointestinal Bleeding; Gastro Intestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This is an obsevational cohort study — no intervention

SUMMARY:
The goal of this study is to identify significant clinical and laboratory risk factors in pediatric patients with significant upper gastrointestinal bleeding. This is defined as bleeding that necessitates an upper endoscopic evaluation to either diagnose or treat upper GI bleeding during their hospital admission. If a predictive/risk stratification relationship exists, these data could permit a more effective triaging and intervention scheme in pediatric patients presenting with complaints of gastrointestinal bleeding. In addition we want to get a better understanding of the re-bleeding rate after endoscopic therapy for upper GI bleeding and if there are any identifiable risk factors for re-bleeding. Lastly we want to understand best practice management for upper GI bleeding.

DETAILED DESCRIPTION:
A. Specific Aims/Objectives:

The goal of this study is to identify significant clinical and laboratory risk factors in pediatric patients with significant upper gastrointestinal bleeding. This is defined as bleeding that necessitates an upper endoscopic evaluation to either diagnose or treat upper GI bleeding during their hospital admission. If a predictive/risk stratification relationship exists, these data could permit a more effective triaging and intervention scheme in pediatric patients presenting with complaints of gastrointestinal bleeding. In addition we want to get a better understanding of the re-bleeding rate after endoscopic therapy for upper GI bleeding and if there are any identifiable risk factors for re-bleeding. Lastly we want to understand best practice management for upper GI bleeding.

B. Background and Significance:

Gastrointestinal (GI) hemorrhage is a potentially life-threatening presentation that the pediatric gastroenterologist must recognize, and manage appropriately. Classification is generally divided between upper or lower GI bleeding, based on the origin of bleeding relative to hemorrhages the Ligament of Treitz. The incidence of GI bleeding in children is not well established in the pediatric population. For upper GI bleeds most large, prospective studies have assessed incidence in pediatric critical care settings. In one prospective study of 984 patients, upper GI bleeds occurred in 6.4% of admissions receiving on prophylactic therapy. Other studies have shown upper GI bleeding in as many as 25% of pediatric intensive care admissions without prophylaxis. There is no data on the incidence of pediatric GI bleeds that requires endoscopic therapy.

Pediatric studies are lacking with respect to risk stratification and decisional algorithms in managing pediatric acute upper gastrointestinal bleeding. Adult literature supports accurate stratification of risk based on clinical history, physical examination, and laboratory measures. Additionally, endoscopic interventions not only allow for therapeutic interventions but also prognosticate based on visual findings. Similar pediatric literature is not available thus giving rise to large amounts of variability both center to center as well as within centers regarding management decision making.

C. Design and Methods:

* Prospective, observational analysis of inpatient and ambulatory records of pediatric patients at Boston Children's Hospital beginning upon IRB approval.
* We will identify pediatric patients </= 21 years old presenting acutely to the emergency room, ambulatory clinic or as current inpatients who require endoscopic evaluation for acute upper gastrointestinal bleed and potential treatment.
* Data collected will include clinical signs and symptoms and physical exam features, laboratory studies and endoscopic findings
* Identified patients will then be followed prospectively for outcomes data collection.
* Data collection will include:

  * Clinical history of bleeding onset, acuity, amount, frequency and prior history of gastrointestinal bleed.
  * Medication history
  * Physical examination data including vital signs (heart rate, blood pressure, and oxygen saturation)
  * Laboratory data including
  * Complete blood count
  * Inflammatory markers (ESR and CRP)
  * Liver panel
  * Complete Metabolic Panel
  * Urinanalysis
  * Endoscopic findings as well as data from interventions (cautery, clips, injections)
  * Medical management decisions (acid suppression therapy, oral intake, frequency of laboratory measurement)
  * Outcome data including re-bleeding rates (with respect to endoscopic intervention), laboratory measures, and length of stay.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients will selected based on signs and symptoms of upper gastrointestinal bleeding and their need to have an upper endoscopy performed.

Exclusion Criteria:

* None

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All pediatric patients who present to the hospital or are currently hospitalized and presented with clinical signs of upper gastric intestinal bleeding that are severe enough that warrant the physician to perform an upper endoscopy.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Develop a predictive/risk stratification algorithm for pediatric upper gastric intestinal bleeding | 3 years
  Identification of prognostic clinical history, physical examination, and laboratory measure risk factors that can predict/risk stratifies significant upper gastrointestinal bleeding in children.

SECONDARY OUTCOMES:
Medical Management Strategies | 3 years
  Identify successful medical management strategies in pediatric patients diagnosed with acute upper gastrointestinal bleed
Endoscopic Management Strategies | 3 years
  Identify successful endoscopic and medical interventions measured by incidence rate of re-bleeding
Re-Bleeding Risk Factors | 3 years
  Identify pre-existing risk factors or clinical factors associated with re-bleeding rates following initial endoscopic or surgical intervention.
Identify Average length of Stay for Upper Gastrointestinal Bleeding | 3 years
  Identify length of medical stabilization and/or observation prior to either endoscopic or surgical intervention measured in hours or days in medical supervision and subsequent outcome, incidence of re-bleeding,
Identify the incidence of significant upper gastrointestinal bleed in all pediatric hospital admission. | 3 years
  Identify the incidence of significant upper gastrointestinal bleed in all pediatric hospital admission.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Manfredi, MD, Principal Investigator — Boston Children's Hospital
Locations (3):
- United States (3):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Childrens Hospital, Boston, Massachusetts
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No